CLINICAL TRIAL: NCT01577589
Title: A Phase I, Single-center, 2-part, Randomized, 2-way Crossover Study to Assess the Local Tolerability and Safety (Multiple-dose) and to Assess the Pharmacokinetics, Safety, and Tolerability (Single-dose) of Ceftaroline in Healthy Subjects When Ceftaroline Fosamil is Diluted in Various Infusion Volume
Brief Title: A 2-part Study to Assess Local Tolerability, Safety and Pharmacokinetics of Ceftaroline in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: D3720C00015
Record Dates: First submitted 2012-04-05; First posted 2012-04-16 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: Phase 1; healthy volunteers; cross-over study; ceftaroline fosamil; various infusion volumes; local tolerability; Cmax; tmax; AUC
MeSH Terms: interventions — Ceftaroline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (6):
- A (Experimental): 600 mg ceftaroline fosamil in 50 ml infusion volume
  Interventions: Drug: 600 mg ceftaroline fosamil in 50 ml infusion volume
- B (Placebo Comparator): Placebo in 50 ml infusion volume
  Interventions: Drug: Placebo in 50 ml infusion volume
- C (Experimental): 600 ceftaroline fosamil in 250 ml infusion volume
  Interventions: Drug: 600 ceftaroline fosamil in 250 ml infusion volume
- D (Placebo Comparator): Placebo in 250 ml infusion volume
  Interventions: Drug: Placebo in 250 ml infusion volume
- E (Experimental): 600 mg ceftaroline in 100 ml infusion volume
  Interventions: Drug: 600 mg ceftaroline in 100 ml infusion volume
- F (Placebo Comparator): Placebo in 100 ml infusion volume
  Interventions: Drug: Placebo in 100 ml infusion volume

INTERVENTIONS:
Drug: 600 mg ceftaroline fosamil in 50 ml infusion volume — IV infusion
  Arms: A
Drug: Placebo in 50 ml infusion volume — IV infusion
  Arms: B
Drug: 600 ceftaroline fosamil in 250 ml infusion volume — IV infusion
  Arms: C
Drug: Placebo in 250 ml infusion volume — IV infusion
  Arms: D
Drug: 600 mg ceftaroline in 100 ml infusion volume — IV infusion
  Arms: E
Drug: Placebo in 100 ml infusion volume — IV infusion
  Arms: F

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of Ceftaroline 600 mg when administered by varying infusion volumes.

DETAILED DESCRIPTION:
A Phase I, Single-center, 2-part, Randomized, 2-way Crossover Study to Assess the Local Tolerability and Safety (Multiple-dose) and to Assess the Pharmacokinetics, Safety, and Tolerability (Single-dose) of Ceftaroline in Healthy Subjects when Ceftaroline Fosamil is Diluted in Various Infusion Volume

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific requirements
* Women of childbearing potential must have a negative pregnancy test, be non-lactating, and be using a highly effective form of birth control for 3 months prior to enrollment, during the study, and for 3 months after completion of all study-related proceed
* Male volunteers must be willing to use barrier contraception from the first day of dosing until 3 months after the last dose of IP.
* Have a body mass index (BMI) between 18 and 30 kg/m2, and weigh at least 50 kg
* Healthy male and/or female volunteers between the ages of 18 to 75 years inclusive, with veins on the back of both hands and both forearms suitable for cannulation or repeated venipuncture.

Exclusion Criteria:

* Use of any other investigational compound or participation in another clinical trial within 1 month prior to first administration of IP in this study
* History of any clinically significant disease or disorder (e.g., neurological, haematological, psychiatric, gastrointestinal, hepatic, renal disease)
* Positive serology result on screening for serum hepatitis B surface antigen, hepatitis C antibody (HCV), or human immunodeficiency virus (HIV)
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
* Any clinically significant abnormalities in the physical examination, lab, 12-lead ECG or vital signs as judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
24-hour pharmacokinetic profile in terms of (see description) for ceftaroline following single-dose administration of ceftaroline fosamil 600 mg diluted in various infusion volumes | Pre-dose, 20 min, 40 min, 60 min, 65 min, 75 min, 90 min, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h, 24 h post-dose
  Maximum plasma concentration (Cmax) Time to maximum concentration (tmax) Area under the concentration-time curve from zero to infinity (AUC) Area under the plasma concentration-time curve from zero to time of the last quantifiable concentrations [AUC(0-t)] Area under the plasma concentration-time curve from zero to 12 hours after the start of the infusion [AUC(0-12)]
24-hour pharmacokinetic profile in terms of (see description)for ceftaroline following single-dose administration of ceftaroline fosamil 600 mg diluted in various infusion volumes | Pre-dose, 20 min, 40 min, 60 min, 65 min, 75 min, 90 min, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h, 24 h post-dose
  Apparent terminal elimination rate constant (Lz) Half-life associated with the terminal slope (t½Lz),mean residence time (MRT) Total body clearance of drug from plasma (CL) Volume of distribution based on the terminal phase(Vz) Volume of distribution at steady state (Vss) Cmax ratios of ceftaroline/ceftaroline fosamil and ceftaroline M-1/ceftaroline (RM/D,Cmax) AUC ratios of ceftaroline/ceftaroline fosamil and ceftaroline M-1/ceftaroline (RM/D,AUC)
Local tolerability in terms of adverse events including local infusion site tolerability for ceftaroline following ceftaroline 600 mg diluted in various infusion volumes every 12 hours for 72 hours | From baseline to 14 days after first dose
  Baseline is defined as - Screening up.

SECONDARY OUTCOMES:
Safety profile in terms of vital signs, ECG, laboratory variables, physical examination for ceftaroline following ceftaroline 600 mg diluted in various infusion volumes every 12 hours for 72 hours | From baseline to 14 days after first dose
  Baseline is defnied as - Screening up
24-hour pharmacokinetic profile in terms of ( see description) for ceftaroline fosamil and ceftaroline M-1following single-dose administration of ceftaroline fosamil 600 mg diluted in various infusion volumes | Pre-dose, 20 min, 40 min, 60 min, 65 min, 75 min, 90 min, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h, 24 h post-dose
  Maximum plasma concentration (Cmax) Time to maximum concentration (tmax) Area under the concentration-time curve from zero to infinity (AUC) Area under the plasma concentration-time curve from zero to time of the last quantifiable concentrations [AUC(0-t)] Area under the plasma concentration-time curve from zero to 12 hours after the start of the infusion [AUC(0-12)]
24-hour pharmacokinetic profile in terms of ( see description) for ceftaroline fosamil and ceftaroline M-1following single-dose administration of ceftaroline fosamil 600 mg diluted in various infusion volumes | Pre-dose, 20 min, 40 min, 60 min, 65 min, 75 min, 90 min, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h, 24 h post-dose
  Apparent terminal elimination rate constant (Lz) Half-life associated with the terminal slope (t½Lz),mean residence time (MRT) Total body clearance of drug from plasma (CL) Volume of distribution based on the terminal phase(Vz) Volume of distribution at steady state (Vss) Cmax ratios of ceftaroline/ceftaroline fosamil and ceftaroline M-1/ceftaroline (RM/D,Cmax) AUC ratios of ceftaroline/ceftaroline fosamil and ceftaroline M-1/ceftaroline (RM/D,AUC)
Safety and tolerability profile in terms of adverse events, vital signs, ECG, laboratory variables, physical exam of ceftaroline following single-dose administration of ceftaroline fosamil 600 mg diluted in various infusion volumes | From baseline to 14 days after first dose)
  Baseline is defined as- Screening up.

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, MD, Study Director — AstraZeneca PharmaceuticalsC2C-7161800 Concord PikePO. Box 15437Wilmington De 19850-5437; Elizabeth Tranter, MBCHB MRCP, Principal Investigator — Hammersmith Medicines Research Cumberland Avenue London NW10 EW UK; Mirjana Kujacic, MD, Study Chair — AstraZeneca Research and DevelopmentSE-431 83 MölndalSweden
Locations (1):
- Research site, London, United Kingdom

REFERENCES:
- [Derived] Edeki T, Kujacic M, Broadhurst H, Li J, Sunzel M. Safety, local tolerability and pharmacokinetics of ceftaroline fosamil administered in a reduced infusion volume. Br J Clin Pharmacol. 2014 Dec;78(6):1291-7. doi: 10.1111/bcp.12465. PMID 25041494
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1378&filename=CSR-D3720C00015.pdf
- See also: CSR-D3720C00015.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1378&filename=CSR-D3720C00015.pdf
- See also: Clinical Study Protocol Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1378&filename=Combined_D3720C00015_Clinical_Study_Protocol_Redacted_V2.pdf